CLINICAL TRIAL: NCT07042048
Title: Placing External Ventricular Drains Using Assistive Augmented Reality or Image-Based Localization: A Randomized Controlled Clinical Trial (PEARL)
Brief Title: Placing External Ventricular Drains Using Assistive Augmented Reality or Image-Based Localization
Acronym: PEARL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cooper Health System (Other)
Responsible Party: Principal Investigator, Corey Mossop, Neurosurgeon, The Cooper Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25-168
Record Dates: First submitted 2025-06-17; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: ICH - Intracerebral Hemorrhage; IVH- Intraventricular Hemorrhage; TBI Traumatic Brain Injury
Keywords: EVD; Augmented Reality; TBI; ICH; Image Guidance
MeSH Terms: conditions — Cerebral Hemorrhage; Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Augmented Reality Assistance (Experimental): Placement of EVDs using augmented reality device
  Interventions: Device: EVD placement - AR assisted
- Stealth Image-guided assistance (Active Comparator): Placement of EVDs using Stealth image-guidance
  Interventions: Device: EVD placement - image-guidance assisted

INTERVENTIONS:
Device: EVD placement - image-guidance assisted — During EVD placement, an image-guided noninvasive systems will be used to assist the operator for EVD catheter tip navigation through a burr hole opening. The use of image-guidance system occurs once during initial EVD placement in this trial.
  Arms: Stealth Image-guided assistance
Device: EVD placement - AR assisted — During EVD placement, an AR system will be used to assist the operator for EVD catheter tip navigation through a burr hole opening. The use of AR occurs once during initial EVD placement in this trial.
  Arms: Augmented Reality Assistance

SUMMARY:
The goal of this clinical trial is to assess if EVD placement using augmented reality is non inferior to image-guidance systems for assistance in adult patients needing an EVD for spontaneous ICH with IVH or severe TBI. The main question it aims to answer is:

Can EVDs be placed successfully with at least equal safety and efficacy using augmented reality devices in comparison to using standard image-guidance techniques?

ELIGIBILITY:
Inclusion Criteria:

* adult patient at time of screening
* diagnosis of spontaneous ICH with IVH with severe TBI
* Meet one or more of the following clinical or radiographic criteria:

Tissue swelling on imaging Dysmorphic ventricles on imaging Midline shift >2mm on imaging Mass effect on imaging Evans Index <0.3 on imaging Glasgow Coma Scale 3-8

* admitted to Cooper University Health
* requires an EVD

Exclusion Criteria:

* Other concomitant intracranial pathology (e.g., tumor, tumor-related edema/hemorrhage, congenital condition, etc.)
* Concurrent participation in another research protocol for investigation of an experimental therapy
* Known or suspected inability to adhere to study protocol or protocol requirements, as per the discretion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Successful EVD catheter placement | During procedure
  Post-procedural non-contrast head CT will be reviewed by masked assessor to evaluate success of EVD placement per the Kakarla grading system. This grading system classifies catheter positioning into three grades based on postoperative imaging. Grade 1 indicates optimal placement in the ipsilateral frontal horn or third ventricle for effective drainage. Grade 2 represents functional but non-ideal placement in the contralateral ventricle or non-eloquent cortex. Grade 3 denotes suboptimal placement in eloquent cortex or non-target spaces, potentially leading to complications. Thus, a higher score means a worse outcome.
rate of complication during placement | During procedure

SECONDARY OUTCOMES:
rate of catheter tip dispositions | During procedure
number of passes for placement | During procedure
rate of AR or Stealth overlay failures on first try | During procedure
rate of EVD failure | from placement to removal of EVD and assessed up to two weeks after
EVD dislodgment of occlusion | from placement to removal of EVD and assessed up to two weeks after
rate of EVD replacement or revision | During procedure
rate of EVD associated hemorrhage | from placement to removal of EVD and assessed up to two weeks after
rate if EVD-associated infection | from placement to removal of EVD and assessed up to two weeks after

CONTACTS AND LOCATIONS:
Locations (1):
- Cooper University Health, Camden, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided